CLINICAL TRIAL: NCT04524013
Title: Swiss National Iodine Survey 2020
Status: Completed | Type: Observational
Sponsor: Isabelle Herter-Aeberli (Other)
Collaborators: Department of Epidemiology and Health Services, Unisanté, Lausanne (Unknown); University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor-Investigator, Isabelle Herter-Aeberli, Senior Scientist, PhD, Swiss Federal Institute of Technology
Organization: Swiss Federal Institute of Technology (Other)
Other Study IDs: 2020-00192
Record Dates: First submitted 2020-08-12; First posted 2020-08-24 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — spot urine samples from women and children, dried blood spots from women.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- School aged children
  Interventions: Other: There is no intervention. It is an observational study.
- Pregnant women
  Interventions: Other: There is no intervention. It is an observational study.

INTERVENTIONS:
Other: There is no intervention. It is an observational study. — There is not intervention

SUMMARY:
This study will assess iodine status in school aged children and pregnant women is Switzerland. In addition, thyroid status and omega-3 index will be assessed in pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* for pregnant women: confirmed pregnancy
* living in Switzerland for min 1 year

Exclusion Criteria:

* no history of major medical illness
* no iodine containing contrast agents or medication in the past 6 months

Ages: 6 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — In the group of pregnant women only pregnant women can participate. The only criteria is that the be pregnant.
Study Population: Both groups: nationally representative sample selected through schools (children) and gynecologists (women).
  School aged children: aged between 6 and 12 years Pregnant women: aged between 18 and 44 years, pregnant
Sampling Method: Probability Sample
Enrollment: 875 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Urinary iodine concentration | Baseline
  urinary iodine concentration in spot urine samples

SECONDARY OUTCOMES:
Urinary creatinine concentration | Baseline
  Urinary creatinine concentration in spot urine samples
Urinary sodium concentration | Baseline
  Urinary sodium concentration in spot urine samples
Urinary fluoride concentration | Baseline
  Urinary fluoride concentration in spot urine samples
Thyroid stimulating hormone | Baseline
  TSH from dried blood spots
T3 | Baseline
  T3 from dried blood spots
T4 | Baseline
  T4 from dried blood spots
Omega 3 index | Baseline
  Omega 3 index from dried blood spots

OTHER OUTCOMES:
Weight | Baseline
Height | Baseline
Omega 3 intake | Baseline
  Assessment of omega 3 intake using a food frequency questionnaire
Depressive symptoms | Baseline
  Assessment of depressive symptoms using the Edinburgh Postnatal Depression Scale (EPDS).

CONTACTS AND LOCATIONS:
Locations (1):
- Human Nutrition Laboratory, ETH Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fischer L, Andersson M, Braegger C, Herter-Aeberli I; Swiss Iodine Study Collaborators. Iodine intake in the Swiss population 100 years after the introduction of iodised salt: a cross-sectional national study in children and pregnant women. Eur J Nutr. 2024 Mar;63(2):573-587. doi: 10.1007/s00394-023-03287-6. Epub 2023 Dec 23. PMID 38141138